CLINICAL TRIAL: NCT05450549
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL919 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL919 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-G-0001; 2022-000756-10 (EudraCT Number)
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DNL919 (Healthy Participant) (Experimental)
  Interventions: Drug: DNL919
- Placebo (Healthy Participant) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL919 — Single doses
  Arms: DNL919 (Healthy Participant)
Drug: Placebo — Single doses
  Arms: Placebo (Healthy Participant)

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled single ascending dose (SAD) study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DNL919.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Female participants of non-childbearing potential (surgically sterilized or post menopausal) or male participants, aged 18 to 55 years, inclusive
* BMI 18.5 to <30 kg/m²
* When engaging in sex with a woman of child bearing potential, both the male participant and his female partner must use highly effective contraception

Key Exclusion Criteria:

* History of clinically significant neurologic, psychiatric, endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematologic, immunologic, or allergic disease, or other major disorders
* History of malignancy
* History of clinically significant stroke
* History of cognitive impairment
* Positive serum pregnancy test at screening, positive urine pregnancy test at baseline visit, or currently lactating or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence, severity, and seriousness of treatment-emergent adverse events (TEAEs) | Up to 45 days

SECONDARY OUTCOMES:
PK Parameter: Maximum concentration (Cmax) of DNL919 in serum | Up to 45 days
PK Parameter: Area under the concentration-time curve from time zero to infinity (AUCinf) | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Claire Meyer, MD, Study Director — Denali Therapeutics Inc.
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shao Q, Chen S, Zheng Y, Xu W, Chen J, Shao W, Wang Q, Li C, Wang X. Crucial role of microglia-mediated myelin sheath damage in vascular dementia: Antecedents and consequences. Neural Regen Res. 2026 Mar 1;21(3):1000-1012. doi: 10.4103/NRR.NRR-D-24-01109. Epub 2025 Mar 25. PMID 40145953